CLINICAL TRIAL: NCT02444000
Title: A Randomized Trial of Delayed Radiotherapy in Patients With Newly Diagnosed 1p/19q Codeleted Anaplastic Oligodendroglial Tumors: the POLCA Trial.
Brief Title: gliomasPCV Only in 1p/19q Codeleted Anaplastic Gliomas
Acronym: POLCA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Association de Neuro-Oncologues d'Expression Francaise (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P130917
Record Dates: First submitted 2015-05-12; First posted 2015-05-14 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Anaplastic Gliomas With 1p/19q Codeletion
Keywords: chemotherapy; PCV; radiotherapy; post operative treatment; anaplastic gliomas; 1p/19q codeletion; cognition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental (Experimental): Administration of 6 cycles of PCV chemotherapy PCV chemotherapy is given as: Day 1: CCNU 110 mg/m2 orally; Days 8 and 29: vincristine 1.4 mg/m2 IV; Days 8 to 21: procarbazine 60 mg/m2 orally
  Interventions: Drug: PCV chemotherapy alone
- control (Active Comparator): radiotherapy followed by 6 cycles of PCV chemotherapy given as: Day 1: CCNU 110 mg/m2 orally; Days 8 and 29: vincristine 1.4 mg/m2 IV; Days 8 to 21: procarbazine 60 mg/m2 orally
  Interventions: Drug: Radiotherapy+PCV chemotherapy

INTERVENTIONS:
Drug: PCV chemotherapy alone — PCV cycles are 6 weeks long
  PCV chemotherapy is given as:
  Day 1: CCNU 110 mg/m2 orally; Days 8 and 29: vincristine 1.4 mg/m2 IV; Days 8 to 21: procarbazine 60 mg/m2 orally
  Arms: experimental
Drug: Radiotherapy+PCV chemotherapy — Radiotherapy followed by 6 cycles of PCV
  Arms: control

SUMMARY:
Patients with 1p/19q-codeleted anaplastic gliomas treated with RT + PCV are at risk of neurocognitive deterioration. Treating these patients with PCV alone (could reduce the risk of neurocognitive deterioration without impairing overall survival.

DETAILED DESCRIPTION:
Multicentric, Randomized phase III study (1:1), Population: newly diagnosed 1p/19-codeleted anaplastic gliomas, Primary objective: To determine whether treating newly diagnosed 1p/19q-codeleted anaplastic gliomas with PCV alone can increase overall survival without neurocognitive deterioration Control group: radiotherapy followed by 6 cycles of PCV chemotherapy. Experimental group: 6 cycles of PCV chemotherapy (radiotherapy being deferred at the time of progression).

Number of centres participating: the 33 centers of the POLA network Recruitment duration: 7 years, the accrual rate being 40 patients per year, and patients are followed-up until the end of the trial.

ELIGIBILITY:
Inclusion criteria :

Histological confirmation of anaplastic glioma by central pathological review

* Tumor is co-deleted for 1p and 19q
* Age ≥ 18 years of age
* Newly diagnosed and ≤3 months from surgical diagnosis
* Willing and able to complete neurocognitive examination and the QOL
* Karnofsky performance status ≥ 60
* The following laboratory values obtained ≤ 21 days prior to registration:
* Absolute neutrophil count (ANC) ≥1500 /mm3
* Platelet count ≥100,000 / mm3
* Hemoglobin > 9.0 g/dL
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
* SGOT (AST) ≤ 3 x ULN
* Negative serum or urine pregnancy test done ≤ 7 days prior to registration, for women of childbearing potential only.
* Provide informed written consent

Exclusion criteria :

* Pregnant and nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception during this study and for up to 6 months following the completion of PCV.
* Received any prior radiation therapy or chemotherapy for any CNS neoplasm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2015-09-22 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2024-09-21 (Actual)

PRIMARY OUTCOMES:
Survival without neurocognitive deterioration | 9 years
  Survival without neurocognitive deterioration (whatever the cause of deterioration, i.e toxicity or tumor progression) defined as the time from study registration to failure in any of the 6 cognitive domains that will be explored (i.e memory, working memory, language, visuo-spatial ability, cognitive executive functions, behavioral executive functions) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
progression free survival | 9 years
overall survival | 9 years

CONTACTS AND LOCATIONS:
Overall Officials: Caroline DEHAIS, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (33):
- France (33):
  - CHU d'Amiens- CHU nord, Amiens
  - CHU D'Anger, Angers
  - CHU annecy genevois, Annecy
  - CHU de Bordaux, Bordeaux
  - Hopital de la Cavale Blanche, Brest
  - CHU de Caen, Caen
  - Hopital Gabriel Montpied, Clermont-Ferrand
  - CH Louis Pasteur, Colmar
  - Hopital François Mitterand, Dijon
  - CHU Sud Réunion, La Réunion
  - Hopital Roger Salengro, Lille
  - Chu Dupuytren, Limoges
  - Centre Hospitalier de Bretagne Sud - Hôpital du Scorff, Lorient
  - GH Est-Institut d'hématologie et d'oncologie pédiatrique IHOP, Lyon
  - Hôpital Pierre Wertheimer, Lyon
  - CHU la Timone, Marseille
  - Hopital CLAIRVAL, Marseille
  - ICM, Institut régional du Cancer de Montpellier, Montpellier
  - Institut de Cancérologie de l'Ouest (ICO) - site CLCC René Gauducheau, Nantes
  - Hopital PASTEUR, Nice
  - HIA du Val de Grâce, Paris
  - Hopital Saint Louis, Paris
  - Groupe Hospitalier Pitié Salpetriere, Paris
  - Centre Hospitalier Perpignan, Perpignan
  - CHU de Poitiers, Poitiers
  - CLCC Eugène Marquis, Rennes
  - CHU de Rouen, Rouen
  - Hôpital Nord, CHU de Saint-Etienne, Saint-Etienne
  - Institut Pul STRAUSS, Strasbourg
  - Hôpital Foch, Suresnes
  - IUCT Oncopole - CLCC Institut Claudius Regaud, Toulouse
  - CHU Bretonneau, Tours
  - CLCC Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No